CLINICAL TRIAL: NCT04420559
Title: The Use of Virtual Reality and Distraction Cards to Reduce Pain During Intramuscular Benzathine Penicillin Injection Procedure in Adults: A Randomized Controlled Trial
Brief Title: Intramuscular Benzathine Penicillin Injection Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Tulay Basak, Head of Fundamentals of Nursing Department, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18/18
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Injection Site Discomfort
MeSH Terms: interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental)
  Interventions: Other: Intramuscular Injection
- Distraction Card (Experimental)
  Interventions: Other: Intramuscular Injection
- Control (No Intervention)

INTERVENTIONS:
Other: Intramuscular Injection — Intramuscular Benzathine Penicillin Injection Procedure
  Arms: Distraction Card; Virtual Reality

SUMMARY:
The aim of this study was the determination of the effect of applying VR and DC distraction methods on patients' pain and satisfaction levels during IM benzathine penicillin injection.

The research hypothesis:

1. Are Virtual Reality and Distraction Card effective in reducing pain due to injection of IM benzathine penicillin?
2. Does the use of Virtual Reality and Distraction Card during the injection process of IM benzathine penicillin have an effect on patient satisfaction?

ELIGIBILITY:
Inclusion Criteria:

* agree to participate in the research,
* being over the age of 18,
* being native speaker,
* not having vision and hearing problems,
* being prescribed benzathine penicillin with a dose of 1.200.000 IU,
* being experienced of IM injection,
* not having IM injection for the last 1 month

Exclusion Criteria:

* volunteers who have scar, incision, lipodystrophy, abscess, necrosis, hematoma, ecchymosis, infection, pain and paralysis at the VG site
* volunteers are excluded if the injection process cannot be performed at one time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 91 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for pain measurement | 4 months
  (Minimum score: 0 ; Maximum score:10) Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Visual Analog Scale for satisfaction measurement (Minimum score: 0 ; Maximum score:10) | 4 months
  (Minimum score: 0 ; Maximum score:10) Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tulay Basak, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basak T, Demirtas A, Yorubulut SM. Virtual reality and distraction cards to reduce pain during intramuscular benzathine penicillin injection procedure in adults: A randomized controlled trial. J Adv Nurs. 2021 May;77(5):2511-2518. doi: 10.1111/jan.14782. Epub 2021 Feb 19. PMID 33608955